CLINICAL TRIAL: NCT03335215
Title: Interest of Cognitive Remediation for the Reduction of Consumption in Alcohol Disorders
Brief Title: Cognitive Remediation in Alcohol Disorders
Acronym: ALCOSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-123
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Alcohol Disorders
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive remediation (Experimental): The innovative nature of this cognitive remediation program is that it integrates both neuropsychological psychoeducation, the principles of reeducation of altered cognitive functions and the setting in addictological context benefiting from the interactions of the group situation. Thus, during the three months of REMED management, six modules corresponding to six altered cognitive domains. The REMED group will benefit from cognitive remediation of episodic memory disorders, executive and attentional functions, and the theory of the mind integrating psychoeducation, training and systematic situations related to an alcoholic context.
  Interventions: Other: cognitive remediation
- usual care (No Intervention)

INTERVENTIONS:
Other: cognitive remediation — The innovative nature of this program is that it integrates both neuropsychological psychoeducation, the principles of reeducation of altered cognitive functions and the setting in addictological context benefiting from the interactions of the group situation. Thus, during the three months of REMED management, six modules corresponding to six altered cognitive domains that may have an impact on the maintenance of the therapeutic contract will be offered to patients. The REMED group will benefit from cognitive remediation of episodic memory disorders, executive and attentional functions, and the theory of the mind integrating psychoeducation, training and systematic situations related to an alcoholic context. The different procedures of neuropsychological management (facilitation, use of preserved capacities and compensation) will help to integrate the concepts and addictological strategies necessary to maintain the therapeutic contract taking into account cognitive impairments.
  Arms: cognitive remediation

SUMMARY:
The individual and societal cost of alcohol use disorders (TUAL), present in 10% of the population in France, is considerable. Despite psychotherapeutic and drug addiction treatment, the relapse rate remains very high, partly because of their very frequent cognitive disorders. In fact, more than 75% of TUAL patients present to varying degrees neuropsychological alterations that are only rarely detected and never treated. However, these cognitive disorders limit the benefit of psychotherapeutic care, reduce compliance with pharmacological treatments and hinder the patient's ability to change his behavior with respect to alcohol. An innovative way to promote the maintenance of the therapeutic contract, and therefore to reduce alcohol consumption in these patients, would be to improve their cognitive functioning. The objective of this study is to measure the efficacy of a non-drug treatment, based on a specific and personalized cognitive remediation program, compared to a standard treatment in Day Hospitalization, in order to reduce the rate of relapse very high in TUAL. It is a randomized, single-blind study with two parallel groups of patients with post-weaning neuropsychological disorders: REMED (cognitive remediation) and CONTROL (usual care).

ELIGIBILITY:
Inclusion Criteria:

* Patient male or female aged 18 to 60, French speaking and affiliated to the social security system
* Patient with TUAL (DSM-5) at the forefront of alcohol use disorders at the time of inclusion
* Patient with neuropsychological disorders objectified on BEARNI (BEARNI for Brief Evaluation of Alcohol-Related Neuropsychological Evaluation, Ritz et al., 2015 cut-off cognitive score = 13, adding a point for patients with bachelor level or lower) and confirmed at the neuropsychological checkup showing pathological performance (at least two free or total recalls of RL / RI 16 <-1.65 and / or RBMT IGM <-1.65 OR number of persecutory or deficit errors at MCST <-1.65 and / or at least two BADS subtests with a score of <or = 2 (except temporal judgment)). Evaluation (BEARNI) at least 48h after stopping benzodiazepines
* Patient weaned of alcohol, that is to say between 5 and 21 days after stopping alcohol, after disappearing signs of withdrawal (Cushman score <2) and stopping benzodiazepines
* First hospitalization type day hospital (not necessarily first weaning)
* Patient having been informed of the study and being able to give written informed consent.

Exclusion Criteria:

* Patient with severe and long-lasting neurological complications related to alcohol (Korsakoff syndrome, fetal alcohol syndrome, ...)
* Patient with a disorder of severe use of another psychoactive substance according to DSM-5, except tobacco
* Patient with motor or sensory deficit making cognitive remediation impossible
* Patient previously included or already included in another biomedical research
* Homeless patient

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
total quantity of alcohol consumed in 3 months (measured in units of pure alcohol, 1 unit = 10g of alcohol). | baseline until 3 month of intervention
  using TimeLine-Follow-Back tracking method (TLFB)

IPD SHARING:
Plan to Share IPD: No